CLINICAL TRIAL: NCT05310708
Title: Validation Study of a Patch-based PSG System
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Onera BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIP_Protocol_Onera_R01
Record Dates: First submitted 2022-01-27; First posted 2022-04-05 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Polysomnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Validation Study of a patch-based PSG system (Experimental): Measuring and recording multiple physiological parameters from a patient which are used by clinicians to make a decision on the diagnosis of sleep.
  Interventions: Diagnostic Test: Polysomnography

INTERVENTIONS:
Diagnostic Test: Polysomnography — Measuring and recording multiple physiological parameters from a patient which are used by clinicians to make a decision on the diagnosis of sleep.

SUMMARY:
This study is a study that qualifies as "other clinical investigation" under Art. 82 MDR and §47 Abs. 3 MPDG with a CE-marked device that aims to demonstrate that the physiological signals from the Onera STS system are substantially equivalent to physiological systems recorded by traditional PSG systems. Furthermore, the study aims to identify the proportion of users who can successfully perform an overnight Onera STS study in an unsupervised home setting. The Onera STS will be used within its approved indication, and the study participants will not be subjected to additional invasive or burdensome procedures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Either referral for a suspected sleep disorder requiring a sleep diagnostic study, or,
* An already diagnosed sleep disorder requiring a planned follow-up PSG.

Exclusion Criteria:

* Inability to provide informed consent
* History of allergic reactions to adhesives or hydrogels or a family history of adhesive skin allergies
* Severe skin condition at sites of patch administration such as wounds, burns or on any damaged skin
* Has an implanted cardiac stimulator or diaphragmatic pacer
* Has an anatomical abnormality that, in the opinion of the Principal Investigator, makes the subject ineligible for inclusion
* Will be exposed to high-frequency surgical equipment, near strong magnetic fields or with devices such as MRIs, external cardiac stimulators during their use of the Onera device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2024-06-21 (Estimated); Study Completion 2024-06-21 (Estimated)

PRIMARY OUTCOMES:
EOG left | 1 year
  Electrooculogram (EOG) is measured on the left side. Here, electrical activity of the eye is measured with an electrode and expressed in microvolt[uV].
EOG right | 1 year
  Electrooculogram (EOG) is measured on the right side. Here, electrical activity of the eye is measured with an electrode and expressed in microvolt[uV].
EEG left | 1 year
  Electroencephalogram (EEG) is measured on the left side. Here, electrical activity of the brain is measured with an electrode and expressed in microvolt[uV].
EEG right | 1 year
  Electroencephalogram (EEG) is measured on the right side. Here, electrical activity of the brain is measured with an electrode and expressed in microvolt[uV].
EMG left | 1 year
  Electromyogram (EMG) is measured on the left side. Here, electrical activity of the muscle is measured with an electrode and expressed in microvolt[uV].
EMG right | 1 year
  Electromyogram (EMG) is measured on the right side. Here, electrical activity of the muscle is measured with an electrode and expressed in microvolt[uV].
SpO2 | 1 year
  Oxygen Saturation (SpO2) is derived from red and infrared Photoplethysmography (PPG) which is measured on the forehead with a reflective pulse oximetry sensor.
ECG | 1 year
  Electrocardiogram (ECG) is measured on the chest. Here, electrical activity of the heart is measured with an electrode and expressed in microvolt[mV].
BioZ Flow | 1 year
  Respiratory Flow (BioZ Flow) is derived from the bioimpedance which is measured on the chest with an electrode (expressed: [a.u.]).
BioZ Effort | 1 year
  Respiratory Effort (BioZ Effort) is derived from the bioimpedance which is measured on the chest with an electrode (expressed: [a.u.]).
Activity | 1 year
  The activity is derived from the accelerometer data of the x, y, and z axis, which is measured on the chest and expressed in the gravitational force equivalent[g].
Snoring | 1 year
  Snoring is measured with the microphone imbedded in the sensor on the chest and expressed in Decibel[dB].
Body Position | 1 year
  The body Position is derived from the accelerometer data of the x, y, and z axis, which is measured on the chest and expressed in degrees[deg].
Nasal Cannula Flow | 1 year
  The Nasal Cannula Flow is measured on the belly using a cannula (expressed: [mmH2O]).
EMG Leg | 1 year
  Electromyogram (EMG) is measured on the lower leg. Here, electrical activity of the muscle is measured with an electrode and expressed in microvolt[mV].

SECONDARY OUTCOMES:
Total Sleep Time | 1 year
  The total time spend asleep expressed in minutes or hours.
Time In Bed | 1 year
  The total time spend in bed expressed in minutes or hours.
SOL | 1 year
  Sleep Onset Latency (SOL) is the length of time that it takes to accomplish the transition from full wakefulness to sleep, expressed in minutes or hours.
Wake Time | 1 year
  The total time spend awake expressed in minutes or hours.
Time in N1 | 1 year
  The total time spend in the N1 sleep stage, expressed in minutes or hours.
Time in N2 | 1 year
  The total time spend in the N2 sleep stage, expressed in minutes or hours.
Time in N3 | 1 year
  The total time spend in the N3 sleep stage, expressed in minutes or hours.
Time in REM | 1 year
  The total time spend in the Rapid Eye Movement (REM) sleep stage, expressed in minutes or hours.
Time in NREM | 1 year
  The total time spend in the Non Rapid Eye Movement (NREM), which contains of the N1, N2, N3 sleep stages, expressed in minutes or hours.
REM | 1 year
  Amount of time spend in the Rapid Eye Movement (REM) sleep stage, expressed in percentage [%].
NREM | 1 year
  Amount of time spend in the Non Rapid Eye Movement (NREM) sleep stage, expressed in percentage [%].
REM Onset Latency | 1 year
  The elapsed time between sleep onset and the onset of the first Rapid Eye Movement (REM) sleep period, expressed in minutes or hours.
WASO | 1 year
  Wake After Sleep Onset (WASO) measures wakefulness, excluding the wakefulness occurring before sleep onset, and is expressed in minutes or hours.
AI | 1 year
  The Arousal Index (AI) divides the total number of arousals by the number of hours of sleep, and therefore is an index for the sleep quality. The lower this amount, the better the outcome.
AHI | 1 year
  The Apnea Hypopnea Index (AHI) is the total amount of apnea or hypopnea event per hour of sleep, and therefore is an index for the severity of sleep apnea. The lower this amount, the better the outcome.
SpO2 | 1 year
  Oxygen Saturation (SpO2) is derived from red and infrared Photoplethysmography (PPG) which is measured on the forehead with a reflective pulse oximetry sensor. This will be expressed in the mean, the minimum, and the maximum.
ODI | 1 year
  The Oxygen Desaturation Index (ODI) is the amount of times per hour of sleep that your blood oxygen level drops by 3% from baseline. The lower this amount the better the outcome.
HR | 1 year
  Heart Rate (HR) is the number of times the heart beats per minute, is derived from the Electrocardiogram (ECG), and expressed in beats per minute[bpm].
Set-up Time PSG (not applicable for application in unsupervised home setting) | 1 year
  Comparison of the setup time (fitting and activation) between the Onera STS system and a traditional Polysomnography (PSG) system.

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Schneider, Principal Investigator — Principal Investigator
Locations (7):
- Germany (7):
  - American Sleep Clinic, Frankfurt, Frankfurt Am Main
  - Schlaf- u. Beatmungszentrum Ulm/Blaubeuren, Blaubeuren Abbey
  - Ruhrlandklinik, Zentrum für Schlaf- und Telemedizin, Essen
  - Evang. Kliniken Essen-Mitte, Essen
  - VAMED Klinik Hagen-Ambrock, Hagen
  - Universitätsklinikum Giessen und Marburg, Marburg
  - Krankenhaus Bethanien, Solingen

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymized datasets and 2D images will be shared with Onera for analysis using secure data transfer. Any images of the facial region will have distinguishing features redacted prior to transfer. Pseudonymized PSG and Onera STS studies (raw and scored) will also be shared with Onera. Following transfer, all study data will be stored on a password protected computer and will only be made available to Onera employees who plan to process it in a way that is compatible with the purposes for which it was collected.

REFERENCES:
- [Derived] Viniol C, Galetke W, Woehrle H, Nilius G, Schobel C, Randerath W, Leiter J, Canisius S, Schneider H. Clinical validation of a wireless patch-based polysomnography system. J Clin Sleep Med. 2025 May 1;21(5):813-823. doi: 10.5664/jcsm.11524. PMID 39773950